CLINICAL TRIAL: NCT03803189
Title: Proactive, Personalized Postpartum Mental Healthcare (P3MH): Designing and Testing an eHealth Intervention to Deliver Proactive, Personalized Postpartum Mental Healthcare for New Parents in Primary Care
Brief Title: Proactive, Personalized Postpartum Mental Healthcare
Acronym: P3MH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Women's College Hospital (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Michael Garron Hospital (Other)
Responsible Party: Principal Investigator, Noah Ivers, Family Physician and Scientist, Women's College Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2018-0099-B; PCG-155463 (Other Grant/Funding Number: Canadian Institutes of Health Research (CIHR))
Record Dates: First submitted 2018-12-25; First posted 2019-01-14 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-10

CONDITIONS: Postpartum Depression; Postpartum Blues; Postpartum Anxiety; Postpartum Mood Disorder
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Intervention Model Description: An independent statistician following a 2:1 ratio to increase opportunities to learn about the intervention processes during this pilot trial will randomly allocate consenting patients at each site following the completion of their baseline survey to intervention or usual care using a computer-generated sequence.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The sequence will be concealed to primary care providers and study staff other than the research coordinator who will apply the allocation. Study staff, including analysts, will also be blind to treatment allocation. Patients and healthcare professionals who may interact with study participants cannot be blinded due to the nature of the intervention, but outcome assessment will be blind.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Personalized eToolkit (Experimental): The intervention arm will receive a personalized eToolkit with community and electronic supports each time they complete a survey, and their PCP will receive supports in the EMR to facilitate postpartum mental healthcare.
  Interventions: Behavioral: Usual care plus eToolkit
- Usual care (No Intervention): The control arm will not receive intervention materials, unless they express suicidality, in which case they will receive a message with supports for suicidality including local emergency departments and crisis lines and an urgent message via EMR and fax will be sent to their PCP. Control arm participants will be asked to complete a baseline e-survey in their third trimester, and a follow-up e-survey 24-weeks after their baby is born.

INTERVENTIONS:
Behavioral: Usual care plus eToolkit — The intervention arm will receive repeated e-surveys via email to collect the Edinburgh Postpartum Depression Scale (EPDS) score at baseline and 2, 4, 6, 8, and 12 weeks. Those with EPDS<10 will be triaged as low risk. Those with EPDS 10-18 (without suicidality) will be triaged as symptomatic for non-urgent clinical assessment with a message delivered via the EMR. Those with EPDS≥19 or suicidality will be triaged as requiring immediate follow-up, with an urgent message to their PCP via EMR, phone (if suicidal) and fax. Prompts in the EMR will enable evidence-based clinical care for PPD and PPA, highlight treatment preferences to support shared decision making, and identify appropriate referrals. Intervention arm participants will receive a personalized eToolkit after the completion of each survey. Patients in the intervention group with symptoms will be invited to a telephone interview at 12 weeks postpartum to describe their experience with the intervention.
  Arms: Personalized eToolkit

SUMMARY:
Mental health symptoms - especially depression and anxiety - are very common in new parents, affecting close to 20% of mothers and at least 10% of fathers. When such symptoms progress to severe levels, they can be more difficult to treat. Early identification of symptoms and prompt treatment are ideal. Despite broad awareness that mental health symptoms in new parents are common, few systems are in place to automatically assess and monitor such symptoms. Evidence-based symptom surveys that can identify parents at risk for postpartum mental health disorders exist, and effective medication and non-medication treatment options are available. Yet, most primary care settings do not have systems in place to ensure that parents with mental health problems (and especially fathers) are identified and treated. This study will use a digital application with a customized website, electronic medical record and email integration to engage parents in assessing their mental health symptoms within weeks of the birth of their new baby. Electronic symptom surveys, sent on behalf of the family doctor, will be used to support proactive, personalized postpartum mental healthcare (P3MH). Responses will be used to enable a tailored care plan for the patient, including advice about options for referrals, treatment, and local community-based psycho-educational and/or social supports. This eHealth intervention includes a web-based application for parents and seamless integration in the EMR, so that when the family doctor sees the patient in clinic, relevant information is ready to be discussed. In this study, a co-design process will be carried with patients and health professionals to refine this eHealth intervention, and determine the usability, user experience, and perceived value of this process in terms of whether it enables mental health symptoms to be caught early and managed in the best way possible for each parent. The procedures will also be piloted for a future large-scale evaluation.

DETAILED DESCRIPTION:
This pilot randomized trial seeks to determine the usability and perceived value of a primary care-based eHealth application that: (1) uses a validated tool (EPDS), to identify and monitor depression and anxiety symptoms in new parents; and (2) collects data on contextual factors and treatment preferences that inform the provision of tailored resources to patients and support the PCP to initiate a tailored treatment pathway. The trial will take place at two sites in the Greater Toronto Area: Women's College Hospital Family Practice Health Centre, and South-East Toronto Family Health Team.

Potential participants (e.g. pregnant women and their partners) will be identified and recruited during pregnancy. Participants will be randomized with an allocation ratio of 2:1 to increase opportunities to learn about the intervention processes. Participants in the intervention arm will complete e-surveys to monitor for symptoms at 2, 4, 6, 8 and 12 weeks postpartum. When symptoms are identified, participants will additionally complete information about contextual factors and treatment preferences. A personalized eToolkit for the patient and clinical decision supports for their primary care provider (PCP) will be produced based on responses to the e-surveys at each time-point. The personalized eToolkit with recommendations for each parent will be generated that includes information about online resources, treatment options, and local, community-based psycho-educational and/or social supports. Participants will be emailed a link to their customized set of resources. The application seamlessly integrates into the primary care electronic medical record (EMR) to provide decision support for the primary care provider, and facilitate shared decision making during the clinical encounter regarding treatment and referral options. Participants will also use the eHealth application to monitor their symptoms over time, alert the primary care team regarding changes, and facilitate timely treatment changes as needs evolve. Participants in the control arm will receive usual care from their primary care provider. If they are flagged as symptomatic at baseline (EPDS>15, PHQ-9 and/or GAD-7 > 10) they will be removed from the study, and provided with electronic resources immediately. A message via EMR will be sent to their PCP, and if suicidality is flagged, their PCP will also receive a message via fax and phone.

ELIGIBILITY:
Inclusion Criteria:

* Biological and non-biological new parents of all sex and gender identities
* Must be able to interact with an eHealth intervention (i.e., have a smartphone, and an active email address)
* Must be rostered to a participating primary care provider who works >1 day per week in the participating clinics and provides comprehensive primary care

Exclusion Criteria:

* History of severe mental illness (e.g. schizophrenia, bipolar disorder), active alcohol or substance use disorder, and/or symptomatic at time of recruitment (i.e., EPDS>15. PHQ-9 and/or GAD-7 >10 or suicidality)
* Pregnant women with active mental illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2019-03-14 (Actual); Primary Completion 2021-04-24 (Actual); Study Completion 2021-04-24 (Actual)

PRIMARY OUTCOMES:
Change in Edinburgh Postpartum Depression Scale (EPDS) Score | Baseline, 12 weeks and 24 weeks postpartum
  The primary outcome will assess intervention effectiveness in terms of improved patient-reported mental health outcomes at 12 and 24 weeks postpartum. Scale range: 0-30; EPDS<10 without suicidality indicates low-risk for postpartum depression and anxiety; EPDS 10-18 without suicidality indicates medium-risk for postpartum depression and anxiety; EPDS>19 and/or suicidality indicates high-risk for postpartum depression and anxiety

SECONDARY OUTCOMES:
Time to treatment initiation | 24 weeks postpartum
  Qualitative self-report questionnaire: what treatments were used by participant

OTHER OUTCOMES:
Perceived value of personalized eToolkit | 12 weeks postpartum
  Qualitative self-report questionnaire: perceived value of the intervention, including whether it was adequately personalized and whether it meets the perceived care needs of mothers and their partners; and barriers and facilitators to implementation of and engagement with the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Noah Ivers, MD, PhD, Principal Investigator — Women's College Hospital
Locations (2):
- Canada (2):
  - South East Toronto Family Health Team, Toronto, Ontario
  - Women's College Hospital Family Practice Health Centre, Toronto, Ontario

REFERENCES:
- [Background] Stewart DE, Vigod S. Postpartum Depression. N Engl J Med. 2016 Dec 1;375(22):2177-2186. doi: 10.1056/NEJMcp1607649. No abstract available. PMID 27959754
- [Background] Dennis CL, Falah-Hassani K, Shiri R. Prevalence of antenatal and postnatal anxiety: systematic review and meta-analysis. Br J Psychiatry. 2017 May;210(5):315-323. doi: 10.1192/bjp.bp.116.187179. Epub 2017 Mar 16. PMID 28302701
- [Background] Falah-Hassani K, Shiri R, Dennis CL. The prevalence of antenatal and postnatal co-morbid anxiety and depression: a meta-analysis. Psychol Med. 2017 Sep;47(12):2041-2053. doi: 10.1017/S0033291717000617. Epub 2017 Apr 17. PMID 28414017
- [Background] Paulson JF, Bazemore SD. Prenatal and postpartum depression in fathers and its association with maternal depression: a meta-analysis. JAMA. 2010 May 19;303(19):1961-9. doi: 10.1001/jama.2010.605. PMID 20483973
- [Background] Field T. Postpartum depression effects on early interactions, parenting, and safety practices: a review. Infant Behav Dev. 2010 Feb;33(1):1-6. doi: 10.1016/j.infbeh.2009.10.005. Epub 2009 Dec 3. PMID 19962196
- [Background] Letourneau N, Tryphonopoulos PD, Duffett-Leger L, Stewart M, Benzies K, Dennis CL, Joschko J. Support intervention needs and preferences of fathers affected by postpartum depression. J Perinat Neonatal Nurs. 2012 Jan-Mar;26(1):69-80. doi: 10.1097/JPN.0b013e318241da87. PMID 22293644
- [Background] Legare F, Witteman HO. Shared decision making: examining key elements and barriers to adoption into routine clinical practice. Health Aff (Millwood). 2013 Feb;32(2):276-84. doi: 10.1377/hlthaff.2012.1078. PMID 23381520
- [Background] O'Connor E, Rossom RC, Henninger M, Groom HC, Burda BU. Primary Care Screening for and Treatment of Depression in Pregnant and Postpartum Women: Evidence Report and Systematic Review for the US Preventive Services Task Force. JAMA. 2016 Jan 26;315(4):388-406. doi: 10.1001/jama.2015.18948. PMID 26813212
- [Background] Kingston D, Austin MP, Veldhuyzen van Zanten S, Harvalik P, Giallo R, McDonald SD, MacQueen G, Vermeyden L, Lasiuk G, Sword W, Biringer A. Pregnant Women's Views on the Feasibility and Acceptability of Web-Based Mental Health E-Screening Versus Paper-Based Screening: A Randomized Controlled Trial. J Med Internet Res. 2017 Apr 7;19(4):e88. doi: 10.2196/jmir.6866. PMID 28389421
- [Background] Gibson J, McKenzie-McHarg K, Shakespeare J, Price J, Gray R. A systematic review of studies validating the Edinburgh Postnatal Depression Scale in antepartum and postpartum women. Acta Psychiatr Scand. 2009 May;119(5):350-64. doi: 10.1111/j.1600-0447.2009.01363.x. Epub 2009 Mar 2. PMID 19298573
- [Background] Matthey S, Fisher J, Rowe H. Using the Edinburgh postnatal depression scale to screen for anxiety disorders: conceptual and methodological considerations. J Affect Disord. 2013 Apr 5;146(2):224-30. doi: 10.1016/j.jad.2012.09.009. Epub 2012 Oct 30. PMID 23116811
- [Background] Matthey S, Barnett B, Kavanagh DJ, Howie P. Validation of the Edinburgh Postnatal Depression Scale for men, and comparison of item endorsement with their partners. J Affect Disord. 2001 May;64(2-3):175-84. doi: 10.1016/s0165-0327(00)00236-6. PMID 11313084
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Eldridge SM, Chan CL, Campbell MJ, Bond CM, Hopewell S, Thabane L, Lancaster GA; PAFS consensus group. CONSORT 2010 statement: extension to randomised pilot and feasibility trials. BMJ. 2016 Oct 24;355:i5239. doi: 10.1136/bmj.i5239. PMID 27777223